CLINICAL TRIAL: NCT07126938
Title: An Observational Study to Facilitate the Development of an Alcohol Impairment Detection Device in Healthy Adult Alcohol Users
Brief Title: Alcohol Impairment Detection in Healthy Adult Users With the Gaize Device
Acronym: AAI
Status: Completed | Type: Observational
Sponsor: Gaize (Industry)
Responsible Party: Sponsor
Other Study IDs: 23-GPHAV-01
Record Dates: First submitted 2025-08-07; First posted 2025-08-17 (Actual); Last update posted 2025-08-26 (Actual); Status verified 2025-08

CONDITIONS: Alcohol Impairment; Nystagmus; Virtual Reality; Lack of Smooth Pursuit; Impairment; Alcohol Intoxication; Intoxication
Keywords: Alcohol; Impairment; Intoxication; Impairment Detection Technology; Alcohol intoxication; Ocular
MeSH Terms: conditions — Nystagmus, Pathologic; Alcoholic Intoxication | interventions — Alcoholic Beverages; Ethanol

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | US Export: No

GROUPS / COHORTS (2):
- experimental: Consumes alcohol
  Interventions: Drug: Alcoholic beverage
- control: Does Not Consume Alcohol

INTERVENTIONS:
Drug: Alcoholic beverage — Participants in the experimental group consumed self-selected amounts of alcohol, monitored by study staff to ensure safety and compliance with protocol guidelines. Participants then filled out the remainder of the general health questionnaire, including how many drinks they consumed, and whether or not they feel too impaired to drive a vehicle or go to work.
  Other Names: Alcohol; Ethanol
  Groups: experimental

SUMMARY:
This study evaluates the effectiveness of the Gaize virtual reality headset as a non-invasive tool for detecting alcohol-related impairment through ophthalmic and neurological indicators. A total of 80 participants, evenly divided into an experimental (alcohol-consuming) and control (non-alcohol consuming) group, underwent baseline and post-consumption ocular assessments using the device. These assessments included: Lack of Smooth Pursuit, Horizontal Gaze Nystagmus at Maximum Deviation, Horizontal Gaze Nystagmus with Onset Prior to 45-Degrees, Vertical Gaze Nystagmus, Lack of Convergence, and Pupillary Rebound Dilation. The Gaize headset measured gaze vector and pupil size at 90 hertz per eye.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged between 21 and 45, having given written informed consent to participate in the research trial and certifying that they do not intend to drive post discharge. We will consider extending the observation period based on individual participants' alcohol consumption.
* Having used alcohol at least one time prior.
* Having experienced impairment too severe to allow for safe operation of a vehicle or work from alcohol use.
* Planning to drink alcohol during their time at the study location.
* Without any history of severe reactions or allergy to alcohol.
* Having access to legal alcohol.
* Normal or corrected to normal vision using either glasses or contact lenses, or surgery.

Exclusion Criteria:

* Enrolled in, or participated in another clinical trial within 30 days before the study
* Having a prosthetic eye, blindness, or vision not corrected to normal.
* Severe reactions or allergy to Alcohol. Participants with a history of severe adverse reactions to alcohol (e.g., allergies, intolerances, or medical conditions worsened by alcohol) are excluded.
* Certain Medical Conditions: Participants with medical conditions or medications that could significantly affect cognitive and motor functions are excluded. A detailed list of such conditions and medications will be provided to potential participants during the screening process.
* Pregnancy: Pregnant individuals will be excluded from the study due to the potential risks associated with alcohol consumption during pregnancy.
* History of Severe Motion Sickness: Participants with a history of severe motion sickness in virtual reality environments may be excluded, as they may not tolerate the virtual reality headset well.
* Individuals who have driven a vehicle (car, truck, bicycle, etc.) to the study location will not be eligible for participation.

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: * Age: Participants ranged from 21 to 45 years old, with an average age of 28.5 years (SD = 6.2).
  * Gender Distribution: The study included 60% male and 40% female participants.
  * Race: The sample was predominantly White (70%), followed by Asian (20%), and Black or other races (10%).
  * Weight: Participant weights ranged from 120 lbs to 250 lbs, with an average weight of 180 lbs (SD = 35 lbs).
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2024-03-21 (Actual); Primary Completion 2024-11-22 (Actual); Study Completion 2024-11-22 (Actual)

PRIMARY OUTCOMES:
Alcohol-Associated Ocular Impairments | 1 hour after alcohol consumption
  Number of participants and measurement of Lack of Smooth Pursuit, Horizontal Gaze Nystagmus at Maximum Deviation, Horizontal Gaze Nystagmus with Onset Prior to 45-Degrees, and Vertical Gaze Nystagmus were evaluated before and after alcohol consumption.

SECONDARY OUTCOMES:
Non-Alcohol Associated Ocular Impairments | 1 hour after Alcohol consumption
  Number of participants and measurement of Lack of Convergence, and Pupillary Rebound Dilation were evaluated before and after alcohol consumption.

CONTACTS AND LOCATIONS:
Locations (1):
- Gaize, Inc., Missoula, Montana, United States

IPD SHARING:
Plan to Share IPD: Undecided